CLINICAL TRIAL: NCT01712620
Title: A Pilot Study of the Effect of Spironolactone Therapy on Exercise Capacity and Endothelial Dysfunction in Pulmonary Arterial Hypertension
Brief Title: Spironolactone for Pulmonary Arterial Hypertension
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); University of Pennsylvania (Other); University of Maryland, Baltimore (Other); Medstar Health Research Institute (Other); New England Medical Center, Tufts University School of Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 120211; 12-CC-0211
Record Dates: First submitted 2012-10-20; First posted 2012-10-23 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2025-11-26

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Magnetic Resonance Imaging
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Spironolactone
  Interventions: Drug: Spironolactone
- Group B (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — Initial dose, 25 mg (pink capsule) orally, daily. If well tolerated at 7-9 wks then increased to 50 mg (brown capsule) daily.
  Arms: Group A
Drug: Placebo — Initial dose, pink sugar capsule, daily. If well tolerated at 7-9 wks then changed to brown sugar capsule, daily.
  Arms: Group B

SUMMARY:
Background:

- High blood pressure in the lungs, known as pulmonary arterial hypertension (PAH), is a rare disorder. In spite of recent advances in treatment, the death rate remains unacceptably high. Lung blood vessel function can be harmed by progressive injuries, such as inflammation, leading to worsening of the disease. A drug called spironolactone has been known to improve blood vessel function and reduce inflammation. Some people with PAH take spironolactone to help treat fluid retention. However, its effect on inflammation and blood vessel function in patients with PAH is not known. Researchers want to see if spironolactone can help these conditions in people with PAH.

Objectives:

- To test the effectiveness of spironolactone in treating pulmonary arterial hypertension.

Eligibility:

- Individuals at least 18 years of age with pulmonary arterial hypertension.

Design:

* This study will last for 24 weeks. Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* Participants will take either spironolactone or a placebo. They will take their study drug or placebo for 7 weeks. Treatment will be monitored with regular blood tests.
* In Week 8, participants who have had no reaction to the treatment will receive a higher dose of the drug or placebo.
* In Week 12, participants will have a study visit with heart and lung function tests. They will also have a 6-minute walk test, and provide blood and urine samples.
* After additional study visits for blood samples, participants will have a final visit in Week 24. The tests from Week 12 will be repeated at this visit.

DETAILED DESCRIPTION:
INTRODUCTION:

Pulmonary arterial hypertension (PAH) is a rare disorder associated with poor survival. Endothelial dysfunction resulting from 1) genetic susceptibility, and 2) a triggering stimulus that initiates pulmonary vascular injury, the two-hit hypothesis, appears to play a central role both in the pathogenesis and progression of PAH. Inflammation appears to drive this dysfunctional endothelial phenotype, propagating cycles of injury and repair in genetically susceptible patients with idiopathic PAH (IPAH) and patients with disease-associated PAH. Therapy targeting pulmonary vascular inflammation to interrupt cycles of injury and repair and thereby delay or prevent RV failure and death has not been tested. Spironolactone, a mineralocorticoid receptor (MR) and androgen receptor (AR) antagonist, has been shown to improve endothelial function and reduce inflammation. Current management of patients with severe PAH and NYHA/WHO class IV symptoms includes use of MR antagonists for their diuretic and natriuretic effects once clinical right heart failure has developed. We hypothesize that initiating therapy with spironolactone at an earlier stage of disease in subjects with PAH could provide additional benefits through anti-inflammatory effects and improvements in pulmonary artery endothelial function.

OBJECTIVES:

Patients with IPAH and disease-associated PAH will be recruited to the NIH and enrolled in a randomized, double blinded, placebo-controlled study of early treatment with spironolactone to investigate its effects on exercise capacity, clinical worsening, and vascular inflammation in vivo.

METHODS:

The total number of PAH subjects enrolled will be up to 70. Subjects will undergo 1) standard clinical examinations including 6-minute walk distance and echocardiography; 2) cardiopulmonary exercise testing; 3) plasma profiling of inflammatory and neurohormonal markers; 4) gene expression profiling of peripheral blood mononuclear cells (PBMCs); and 5) high-resolution MRI-based determination of pulmonary vascular and RV structure and function. Safety and tolerability of spironolactone in PAH will be assessed with periodic monitoring for hyperkalemia and renal insufficiency as well as the incidence of drug discontinuation for untoward effects.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. WHO Group 1 PH patients on either no medical therapy or stable medical therapy for at least the past 4 weeks (defined as no new PAH-specific therapy, no change in the dose of current PAH-specific therapy and no change in NYHA/WHO functional classification within the past 4 weeks) are eligible. The following parameters on RHC are required to meet the hemodynamic definition of PAH:

  <!-- -->

  1. mean pulmonary artery pressure of > 25 mmHg at rest,
  2. pulmonary capillary wedge pressure of less than or equal to 15 mmHg (or a left ventricular end-diastolic pressure of less than or equal to 12 mmHg) and
  3. pulmonary vascular resistance of > 3 Wood units (240 dyn.s.cm^-5).

If clinically indicated at the time of enrollment, then a RHC will be performed at the NIH Clinical Center upon study entry under a procedural consent.

2) Females who are able to become pregnant (i.e., are not postmenopausal, have not undergone surgical sterilization, and are sexually active with men) must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to and for the duration of study participation.

EXCLUSION CRITERIA:

1. Patients with WHO Group 1 PH and evidence of right heart failure as defined by:

   1. NYHA/WHO class IV symptoms and
   2. Echocardiographic evidence of severe RV dysfunction and
   3. Clinical evidence of right heart failure which may include, but is not limited to elevated jugular venous pressure, ascites, and lower extremity edema
2. Patients with WHO Group 1 pulmonary hypertension and a prior diagnosis of cirrhosis with portal hypertension as evidenced by a history of ascites, hepatic encephalopathy and/or varices prior to enrollment
3. Patients with WHO Group 1 pulmonary hypertension and evidence of active infection, (HIV patients with two consecutive viral loads of < 500 on their most recent determinations within the past 12 months will be considered to have inactive infection)
4. Patients with WHO Group 1 pulmonary hypertension who have taken spironolactone or eplerenone within the last 30 days
5. Known or suspected allergy to spironolactone
6. Pregnant or breastfeeding women (all women of childbearing potential will be required to have a screening urine or blood pregnancy test)
7. Age <18 years
8. Inability to provide informed written consent for participation in the study
9. Chronic kidney disease (an estimated glomerular filtration rate of < 35 mL/min/1.73m^2 of body surface area)
10. Serum potassium at the time of enrollment of > 5 mEq/L
11. Concurrent use of an ACE inhibitor and angiotensin II receptor blocker

    OR

    Patients currently taking the maximum recommended dose of an ACE inhibitor or an angiotensin II receptor blocker [For patients taking one of these medicines (ACE-Inhibitors or ARBs), the investigators agree to do due diligence by consulting a clinical center pharmacist and/or a standard pharmacy reference (i.e. Micromedex) to certify whether or not the patient is on a maximum dose of the drug.]
12. Women currently taking drospirenone-containing oral contraceptives

The estimated glomerular filtration rate (eGFR) will be calculated using the IDMS-traceable Modification of Diet in Renal Disease (MDRD) equation and corrected for body surface area.

eGFR = 175 x (serum creatinine in mg/dL)^-1.154 x (age in years)^-0.203 x [1.212 if African-American] x [0.742 if female]

(http://www.nkdep.nih.gov/professionals/gfr_calculators/idms_con.htm)

Exclusion Criteria for MRI

These contraindications include but are not limited to the following devices or conditions:

1. Implanted cardiac pacemaker or defibrillator
2. Cochlear Implants
3. Ocular foreign body (e.g. metal shavings)
4. Embedded shrapnel fragments
5. Central nervous system aneurysm clips
6. Implanted neural stimulator
7. Any implanted device that is incompatible with MRI
8. Unsatisfactory performance status as judged by the referring physician such that the subject could not tolerate an MRI scan. Examples of medical conditions that would not be accepted would include unstable angina and severe dyspnea at rest
9. Subjects requiring monitored sedation for MRI studies
10. Subjects with a condition precluding entry into the scanner (e.g. morbid obesity, claustrophobia, etc.)
11. Subjects with severe back-pain or motion disorders who will be unable to tolerate supine positioning within the MRI scanner and hold still for the duration of the examination.

EXCLUSION CRITERIA FOR GADOLINIUM BASED MRI STUDIES ONLY:

1. History of severe allergic reaction to gadolinium contrast agents despite pre- medication with diphenhydramine and prednisone
2. Chronic kidney disease (an estimated glomerular filtration rate of < 60 mL/min/1.73m^2 of body surface area)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2014-01-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in placebo corrected 6-minute walk distance | 6 months
  Change in placebo corrected 6-minute walk distance.

SECONDARY OUTCOMES:
Change in placebo corrected VO2 max | 6 months
Change in right ventricular function | 6 months
Biomarkers of vascular inflammation | 6 months
Rate of study drug discontinuation due to hyperkalemia, renal insufficiency, or other side effects such as breast pain and gynecomastia | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Solomon, M.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Elinoff JM, Rame JE, Forfia PR, Hall MK, Sun J, Gharib AM, Abd-Elmoniem K, Graninger G, Harper B, Danner RL, Solomon MA. A pilot study of the effect of spironolactone therapy on exercise capacity and endothelial dysfunction in pulmonary arterial hypertension: study protocol for a randomized controlled trial. Trials. 2013 Apr 2;14:91. doi: 10.1186/1745-6215-14-91. PMID 23547564
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2012-CC-0211.html